CLINICAL TRIAL: NCT02621645
Title: Early Versus Late Intervention for Twin Reversed Arterial Perfusion Sequence: an Open-label Randomized Controlled Trial: TRAPIST - TRAP Intervention STudy
Brief Title: TRAP Intervention STudy: Early Versus Late Intervention for Twin Reversed Arterial Perfusion Sequence
Acronym: TRAPIST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: St. George's Hospital, University of London (UK sponsor) (Unknown); Leiden University Medical Center (Other); Ospedalo Maggiore Policlinico di Milano, Italy (Unknown); Hospital Universitari Vall d'hebron Barcelona, Spain (Unknown); Centro Médico-Chirurgical et Obstétrical (CMCO) Schiltigheim, France (Unknown); Universitätsklinik für Frauenheilkunde und Geburtshilfe Graz, Austria (Unknown); Ospedale dei Bambini "Vittore Buzzi" Milano, Italy (Unknown); Birmingham Women's Hospital, UK (Unknown); Sheba Medical Center (Other Government); Children's Memorial Hermann Hospital Houston Texas, USA (Unknown); Universitätsklinikum Hamburg-Eppendorf, Germany (Unknown); Mount Sinai Hospital, Canada (Other); University of Pittsburgh (Other); University Hospital Innsbruck, Austria (Unknown); Spedali Civili, University of Brescia, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S58224
Record Dates: First submitted 2015-11-12; First posted 2015-12-03 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Twin Reversal Arterial Perfusion Syndrome
Keywords: monochorionic; TRAP; acardiac twin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early intervention (Experimental): Intervention between 12.0 and 14.0 weeks. Early selective reduction of TRAP mass.
  Interventions: Procedure: Early selective reduction of TRAP mass; Device: Ultrasound-guided intrafetal ablation using a 18 to 20 Gauge needle
- Late intervention (Active Comparator): Intervention between 16.0 and 19.0 weeks. Late selective reduction of TRAP mass. This is the standard timing of the intervention. One of two possible techniques for late reduction is chosen by the treating physician.
  Interventions: Procedure: Late selective reduction of TRAP mass; Device: Ultrasound-guided intrafetal ablation using a 17 to 20 Gauge needle; Device: Laser coagulation of the cord or anastomising vessels through a 17 Gauge to 7 French trocar, with a 1-1,3 mm fetoscope and a 400 µm laser fiber

INTERVENTIONS:
Procedure: Early selective reduction of TRAP mass — Ultrasound-guided intrafetal ablation using an 18 Gauge to 20 Gauge needle
  Arms: Early intervention
Procedure: Late selective reduction of TRAP mass — Ultrasound-guided intrafetal ablation using a 17 Gauge to 20 Gauge needle OR fetoscopic laser coagulation of the cord or anastomising vessels through a 17 Gauge to 7 French trocar, with a 1-1,3 mm fetoscope and a 400 µm laser fiber. The treating physician can decide which technique will be used for the selective reduction.
  Arms: Late intervention
Device: Ultrasound-guided intrafetal ablation using a 18 to 20 Gauge needle
  Arms: Early intervention
Device: Ultrasound-guided intrafetal ablation using a 17 to 20 Gauge needle
  Arms: Late intervention
Device: Laser coagulation of the cord or anastomising vessels through a 17 Gauge to 7 French trocar, with a 1-1,3 mm fetoscope and a 400 µm laser fiber
  Arms: Late intervention

SUMMARY:
Multi-center open-label randomized controlled trial to assess if early intervention (12.0-14.0 weeks) (study group) improves the outcome of TRAP sequence as compared to late intervention (16.0-19.0 weeks) (control group). The investigators will randomly assign women diagnosed with TRAP sequence diagnosed between 12.0 and 13.6 weeks to an early or late intervention group (1:1), using a web-based application and a computer-generated list with random permuted blocks of sizes 2 or 4 (www.sealedenvelope.com), stratified by gestational age (GA) at inclusion (11.6 -12.6 weeks versus 13.0-13.6 weeks). Analysis will be by intention to treat.

DETAILED DESCRIPTION:
The investigators propose to conduct a multi-center open-label randomized controlled trial to assess if early intervention (12.0-14.0 weeks) (study group) improves the outcome of TRAP sequence as compared to late intervention (16.0-19.0 weeks) (control group). The investigators will randomly assign women diagnosed with TRAP sequence diagnosed between 11.6 and 13.6 weeks (1:1) to an early or late intervention group, using a web-based application (www.sealedenvelope.com) with a computer-generated list with random permuted blocks of sizes 2 or 4, stratified by gestational age at inclusion (11.6 -12.6 weeks versus 13.0-13.6 weeks). Analysis will be by intention-to-treat. Outcome will be adjudicated blinded to group allocation.

All interventions will be done under local anaesthesia and/or conscious sedation in sterile conditions by an experienced operator. They must be performed within 1 week after randomisation and at the latest at 14.0 weeks in the early group and 19.0 weeks in the late group. In the early group, only intrafetal coagulation will be used. Intrafetal ablation will be performed under ultrasound guidance using an 18-gauge (1.27 mm) to 20-gauge (0.91 mm) needle with a free-hand technique. The needle is introduced into the pelvis/abdomen of the TRAP mass close to the intra-abdominal portion of the feeding vessel, while avoiding puncture of the placenta and pump twin sac. The procedure is considered successful when there is complete cessation of reverse flow into the TRAP mass on intraoperative color-flow mapping.

In the late intervention/control group either intrafetal coagulation or fetoscopic laser coagulation will be performed of the cord and/or anastomosing vessels, unless the flow has stopped spontaneously or demise of the pump twin has occurred in the meantime. Intrafetal coagulation is done as described above by using a 17-gauge (1.47 mm) to 20-gauge needle. Alternatively, fetoscopic laser coagulation of the cord or anastomosing vessels can be performed through a 17-gauge to 7 French trocar with 1-1,3 mm fetoscope and 400 μm laser fiber. The rationale not to standardize the technique in the late intervention group is that several techniques have been reported for treatment after 16 weeks without any significant differences in outcome. Also, it is usual for the surgeon to adapt the technique to the requirements of each individual case, e.g. for a posterior placenta, the surgeon may prefer fetoscopic rather than intrafetal coagulation. Not restricting the technique to only 1 option will therefore more truly represent current practice and increase the generalizability of the trial's findings.

Patients will be discharged the same day or 1 day after the procedure. Management and follow-up will be similar for the study and the control or current practice group. A follow-up scan is usually performed 1 week after the intervention to check for fetal well-being and exclude anemia. A detailed ultrasound scan will be arranged in a fetal medicine center at 20 and 30 weeks to assess the heart and brain anatomy. Some centers may offer an MRI scan at around 30 weeks as part of the protocol for monochorionic twin pregnancies that underwent an intrauterine intervention. Antenatal, peripartum and postnatal care of the mother will be similar to that of a singleton pregnancy and at the discretion of the referring physician. Intrauterine intervention for TRAP sequence is not an indication for cesarean or elective preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* TRAP sequence in a monochorionic diamniotic twin pregnancy diagnosed between 11.6 and 13.6 weeks, as determined by the crown-rump length of the pump twin in spontaneous conceptions and by the date of insemination or embryonic age at replacement in pregnancies resulting from subfertility treatment
* Women aged 18 years or more, who are able to consent
* Anatomically normal pump twin
* Provide written informed consent to participate in this randomized controlled trial, forms being approved by the Ethical Committees

Exclusion Criteria:

* Contraindication for an intervention due to a severe maternal medical condition or threatening miscarriage
* Inaccessibility of the acardiac twin due to a retroverted uterus, severe maternal obesity, uterine fibroids, bowel or placental superposition
* A major anomaly in the pump twin, requiring surgery or leading to infant death or severe handicap
* Spontaneous arrest of the reverse flow and/or pump twin demise at diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with neonatal survival and birth at or after 34.0 weeks of the pump twin | 2 weeks after expected date of birth

SECONDARY OUTCOMES:
Number of patients with need for re-intervention | 2 weeks after expected date of birth
  This means any kind of fetal intervention, such as repeated intrafetal coagulation, intra-uterine transfusion cord-occlusion...
Number of patients with maternal morbidity | 2 weeks after expected date of birth
  Maternal morbidity is defined as presence of one or more of the following events:
  * Need for transfusion for hemorrhage
  * Abruption
  * Chorioamnionitis as defined on pathology
  * Sepsis
  * Bowel perforation
  * Other serious maternal morbidity requiring admission to ICU
Number of patients with miscarriage | 2 weeks after expected date of birth
  Number of patients with miscarriage before 24 weeks
Number of patients with preterm prelabor rupture of membranes (PPROM) | 2 weeks after expected date of birth
  Number of patients with rupture of membranes before onset of labor and before 37 weeks
Number of patients with preterm birth prior to 28 weeks | 2 weeks after expected date of birth
  Number of patients delivering before 28 weeks
Number of patients with preterm birth prior to 32 weeks | 2 weeks after expected date of birth
  Number of patients delivering before 32 weeks
Number of patients with preterm birth prior to 37 weeks | 2 weeks after expected date of birth
  Number of patients delivering before 37 weeks
Time from randomization to delivery | 2 weeks after expected date of birth
  Number of weeks between randomization and the time of delivery
Time from randomization to PPROM | 2 weeks after expected date of birth
  Number of weeks between randomization and rupture of membranes in patients with PPROM
Birth weight in grams | 42 days (28 days neonatal period+2 weeks postdates) after expected date of birth
Number of patients with stillbirth | 42 days (28 days neonatal period+2 weeks postdates) after expected date of birth
  Stillbirth refers to all patients with antepartum or intrapartum demise of the fetus
Number of patients with neonatal death | 42 days (28 days neonatal period+2 weeks postdates) after expected date of birth
  Demise of a live-born child within the first 28 days of life
Number of patients with severe neonatal morbidity | 42 days (28 days neonatal period+2 weeks postdates) after expected date of birth
  Severe neonatal morbidity is defined as the presence of at least one of the following:
  * chronic lung disease (defined as oxygen dependency at 36 weeks gestational age)
  * patent ductus arteriosus needing medical therapy or surgical closure
  * necrotizing enterocolitis stage 2 or higher
  * retinopathy of prematurity stage 3 or higher
  * ischemic limb injury
  * amniotic band syndrome
  * severe cerebral injury (includes at least one of the following: intraventricular hemorrhage grade 3 or higher, cystic periventricular leukomalacia grade 2 or higher, ventricular dilatation greater than the 97th centile, porencephalic or parenchymal cysts or other severe cerebral lesions).
High volume vs low volume centers of neonatal survival and birth at or after 34.0 weeks of the pump twin and maternal morbidity parameters | 2 weeks after expected date of birth
Number of patients with intact survival rate | 2 years after expected date of birth
  Intact survival rate defined as the number of surviving infants with normal development at two years corrected for prematurity as assessed by the ASQ® score for infant development (Ages & Stages Questionnaire). A score of more than 2 standard deviations below the mean score for term-born children will be considered abnormal.
Number of patients with normal Bayley III score | 2 years after expected date of birth
  Number of patients with normal Bayley III score at two years of age corrected for prematurity

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth Lewi, MD PhD, Study Chair — UZ Leuven
Locations (14):
- Children's Memorial Hermann Hospital, Houston, Texas, United States
- Universitätsklinik für Frauenheilkunde und Geburtshilfe, Graz, Austria
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Mount Sinai Hospital, Toronto, Canada
- Centre Médico-Chirurgical et Obstétrical, Schiltigheim, France
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany
- Sheba Medical Center, Tel Litwinsky, Israel
- Italy (2):
  - Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan
  - Ospedale dei Bambini Vittore Buzzi, Milan
- Leiden University Medical Center, Leiden, Netherlands
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- United Kingdom (3):
  - Birmingham Women's Hospital, Birmingham
  - King's College, London
  - St. George's Hospital, University of London (UK sponsor), London

REFERENCES:
- [Background] Moore TR, Gale S, Benirschke K. Perinatal outcome of forty-nine pregnancies complicated by acardiac twinning. Am J Obstet Gynecol. 1990 Sep;163(3):907-12. doi: 10.1016/0002-9378(90)91094-s. PMID 2206078
- [Background] Pagani G, D'Antonio F, Khalil A, Papageorghiou A, Bhide A, Thilaganathan B. Intrafetal laser treatment for twin reversed arterial perfusion sequence: cohort study and meta-analysis. Ultrasound Obstet Gynecol. 2013 Jul;42(1):6-14. doi: 10.1002/uog.12495. PMID 23640771
- [Background] Hecher K, Lewi L, Gratacos E, Huber A, Ville Y, Deprest J. Twin reversed arterial perfusion: fetoscopic laser coagulation of placental anastomoses or the umbilical cord. Ultrasound Obstet Gynecol. 2006 Oct;28(5):688-91. doi: 10.1002/uog.3816. PMID 16958150
- [Background] Chaveeva P, Poon LC, Sotiriadis A, Kosinski P, Nicolaides KH. Optimal method and timing of intrauterine intervention in twin reversed arterial perfusion sequence: case study and meta-analysis. Fetal Diagn Ther. 2014;35(4):267-79. doi: 10.1159/000358593. Epub 2014 Apr 16. PMID 24751835
- [Background] Lewi L, Valencia C, Gonzalez E, Deprest J, Nicolaides KH. The outcome of twin reversed arterial perfusion sequence diagnosed in the first trimester. Am J Obstet Gynecol. 2010 Sep;203(3):213.e1-4. doi: 10.1016/j.ajog.2010.04.018. Epub 2010 Jun 3. PMID 20522408
- [Background] O'Donoghue K, Barigye O, Pasquini L, Chappell L, Wimalasundera RC, Fisk NM. Interstitial laser therapy for fetal reduction in monochorionic multiple pregnancy: loss rate and association with aplasia cutis congenita. Prenat Diagn. 2008 Jun;28(6):535-43. doi: 10.1002/pd.2025. PMID 18509857
- [Background] Scheier M, Molina FS. Outcome of twin reversed arterial perfusion sequence following treatment with interstitial laser: a retrospective study. Fetal Diagn Ther. 2012;31(1):35-41. doi: 10.1159/000334156. Epub 2011 Dec 23. PMID 22204966
- [Background] Berg C, Holst D, Mallmann MR, Gottschalk I, Gembruch U, Geipel A. Early vs late intervention in twin reversed arterial perfusion sequence. Ultrasound Obstet Gynecol. 2014 Jan;43(1):60-4. doi: 10.1002/uog.12578. PMID 23908075
- [Background] Jelin E, Hirose S, Rand L, Curran P, Feldstein V, Guevara-Gallardo S, Jelin A, Gonzales K, Goldstein R, Lee H. Perinatal outcome of conservative management versus fetal intervention for twin reversed arterial perfusion sequence with a small acardiac twin. Fetal Diagn Ther. 2010;27(3):138-41. doi: 10.1159/000295176. Epub 2010 Mar 9. PMID 20215730
- [Background] Lewi L, Gratacos E, Ortibus E, Van Schoubroeck D, Carreras E, Higueras T, Perapoch J, Deprest J. Pregnancy and infant outcome of 80 consecutive cord coagulations in complicated monochorionic multiple pregnancies. Am J Obstet Gynecol. 2006 Mar;194(3):782-9. doi: 10.1016/j.ajog.2005.09.013. PMID 16522413
- [Background] Kerstjens JM, Nijhuis A, Hulzebos CV, van Imhoff DE, van Wassenaer-Leemhuis AG, van Haastert IC, Lopriore E, Katgert T, Swarte RM, van Lingen RA, Mulder TL, Laarman CR, Steiner K, Dijk PH. The Ages and Stages Questionnaire and Neurodevelopmental Impairment in Two-Year-Old Preterm-Born Children. PLoS One. 2015 Jul 20;10(7):e0133087. doi: 10.1371/journal.pone.0133087. eCollection 2015. PMID 26193474